CLINICAL TRIAL: NCT00207948
Title: Optimizing Antiretroviral Therapy in HIV-Infected Children and Adolescents
Status: Terminated | Type: Observational
Why Stopped: no measurable response was detected at the 50% increase threshold.
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Natella Rakhmanina, MD, Children's National Research Institute
Other Study IDs: 1K12RR017613-03 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus; Protease Inhibitors; Pharmacogenetics; Genes, MDR1, Cytochrome P-450 enzymes; Pharmacokinetics; Pediatrics; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Therapeutic Dose Adjustment: To adjust the doses of medications to meet target therapeutic concentrations
  Interventions: Drug: Dose adjustment of Kaletra

INTERVENTIONS:
Drug: Dose adjustment of Kaletra — Adjust the dose by up to +50% of reccomended dosa off the drug to meet target therapeutic concentrations
  Other Names: Lopinavir; Ritonavir

SUMMARY:
This was a feasibility study aimed at elevating protease inhibitors (PI) dosage as a part of active antiretroviral therapy (HAART). After the pharmacokinetics for the currently prescribed PI were determined,patients with a vIQ<1 were eligible for a 50% dose increase for an 8 week time frame after which their vIQ would be reassessed to determine if increasing their PI dosage thereby increasing the bioavaiability would reduce their viral load.

DETAILED DESCRIPTION:
Although, the use of protease inhibitors (PI) containing highly active antiretroviral therapy (HAART) has led to a remarkable improvement in the prognosis and outcome of HIV infection, only 45% to 70% of treatment-naïve patients who commence HAART achieve complete virological suppression. The emergence of HIV resistance to antiretroviral drugs is one of the main obstacles to the successful long-term suppression of HIV replication. Poor adherence and unfavorable pharmacokinetics (PK) caused by altered absorption, genetic variations in metabolism and drug-drug interactions frequently lead to antiretroviral drug concentrations below the inhibitory concentration for 50% of the viral quasispecies (IC50) and loss of viral suppression.

Enzymes of the cytochrome (CYP) P450 (CYP2C19, CYP3A4, CYP3A5) family located in the liver and small intestine are responsible for the metabolism of PIs. The absence of expression of certain enzymes from this family was recently correlated with a genetic polymorphism, which may have a major role in variation of cytochrome P450-mediated drug metabolism. Results of these studies suggest significant differences in the distribution of the polymorphism associated alleles between ethnic groups, in particular between Caucasians and African Americans. Detection of cytochrome P450 variant alleles and more detailed data on their allelic frequency in various ethnic groups is critical to assess their impact on PK of antiretroviral agents, in particular PIs.

This research proposal is aimed at the development of a novel multidisciplinary approach to optimize HAART in HIV infected children. It is increasingly clear that inter-individual variation in drug metabolism and responsiveness has a strong genetic component. The metabolic pathways leading to drug clearance, bio-availability, and cellular responses are complex, and only beginning to be understood. Key to our understanding of inter-individual responses is identification of the genetic polymorphisms that contribute to this variability, the relative contribution of different genes/SNPs, and the possible interactions between the corresponding protein products or pathways. We propose to develop a dosing regimen of PIs in HIV-infected children that takes into account genetic variability in drug metabolism and transport, and resistance of the dominant viral strain (as determined by virtual phenotype).

In order to do so, the protocol address the following Specific Aims:

* Specific Aim 1 (completed previously): Determine the prevalence of genetic variations in CYP2C19, CYP3A4, CYP3A5, and MDR-1 genes in a cohort of children and adolescents with HIV infection.
* Specific Aim 2 (completed previously): Evaluate the relationship of this genetic variability to the pharmacokinetic parameters (Cmin, Cmax, AUC) and toxicity (graded by the Division of AIDS [DAIDS] classification) of protease inhibitors in pediatric patients with HIV infection.
* Specific Aim 3 (THIS STUDY): Evaluate the impact of dose adjustment of protease inhibitors based on pharmacogenetic profile and virtual inhibitory quotient (VIQ) on clinical outcome (measured by HIV-RNA viral load and CD4+ cell count changes) and toxicity (graded by the DAIDS classification) in pediatric patients with HIV infection.

ELIGIBILITY:
Inclusion criteria:

* Evidence of HIV infection confirmed by positive culture or PCR on at least two occasions, or a positive ELISA and a confirmatory Western Blot. At least one of these tests must be done in an ACTG certified laboratory which is approved to perform the assay for protocol testing
* Age 4-21 years
* Current use of HAART regimen (NRTI or/and NNRTI based) containing a PI
* HIV-RNA levels above 1,000 copies/mL (Stage II)
* vIQ<1 for Kaletra
* Signed informed consent and, if indicated, signed informed assent or waiver of assent.

Exclusion criteria:

* Grade 3-4 DAIDS defined toxicity
* Use of cimetidine (used as the internal standard for the HPLC-MS/MS assay)
* Any active opportunistic infection
* Any of the following laboratory findings at entry: absolute neutrophil count <750 cells/mm3; platelet count <75,000 cells/mm3; AST >3 times upper limit of age adjusted normal values; ALT >3 times upper limit of age adjusted normal values; serum creatinine >1.2mg/dL.
* Patients on dual PI regimen (except when second PI is given for boosting) at the time of enrollment

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The total number of recruited subjects in a previous the study was 78 with 50 subjects on LPV/RTV based ART. Based on PK analysis 4 patients fit inclusion criteria for a dose adjustment feasibility pilot (this study)
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
evaluation of vIQ | 8 weeks
  vIQ would be reassessed to determine if increasing their PI dosage thereby increasing the bioavaiability would reduce their viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Natella Y Rakhmanina, MD, Principal Investigator — Children's National Medical Center, Children's Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Rakhmanina N, van den Anker J, Baghdassarian A, Soldin S, Williams K, Neely MN. Population pharmacokinetics of lopinavir predict suboptimal therapeutic concentrations in treatment-experienced human immunodeficiency virus-infected children. Antimicrob Agents Chemother. 2009 Jun;53(6):2532-8. doi: 10.1128/AAC.01374-08. Epub 2009 Mar 2. PMID 19258274
- [Result] Neely MN, Rakhmanina NY. Comment on: Pharmacokinetics and 48 week efficacy of low-dose lopinavir/ritonavir in HIV-infected children. J Antimicrob Chemother. 2010 Apr;65(4):808-9; author reply 809-10. doi: 10.1093/jac/dkp489. Epub 2010 Jan 19. No abstract available. PMID 20086000
- [Result] Rakhmanina NY, Neely MN, Van Schaik RH, Gordish-Dressman HA, Williams KD, Soldin SJ, van den Anker JN. CYP3A5, ABCB1, and SLCO1B1 polymorphisms and pharmacokinetics and virologic outcome of lopinavir/ritonavir in HIV-infected children. Ther Drug Monit. 2011 Aug;33(4):417-24. doi: 10.1097/FTD.0b013e318225384f. PMID 21743379